CLINICAL TRIAL: NCT05671068
Title: CEREBELLAR INVOLVEMENT IN MOTOR, COGNITIVE AND EMOTIONAL PROCESSES IN MYOCLONUS DYSTONIA
Brief Title: EMOTION & COGNITION IN MYOCLONUS DYSTONIA (AGENT10-ECODYST)
Status: Completed | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: C22-18; 2022-A00786-37 (Other: ID RCB)
Record Dates: First submitted 2022-12-16; First posted 2023-01-04 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Myoclonus-Dystonia; DYT11
MeSH Terms: conditions — Myoclonic dystonia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- DYT-SGCE: Patients with myoclonus dystonia (DYT-SGCE)
- Healthy volunteers: Control group

SUMMARY:
Background:

Myoclonus dystonia (DYT-SGCE) is characterized by myoclonus and dystonia. Such condition is associated with a high prevalence of psychiatric symptoms which are part of the phenotype. The mechanisms underlying these non-motor symptoms are still poorly understood.

Objective:

To investigate the neural correlates of cognition and emotion in DYT-SGCE.

Design:

Participants will have 1 - 2 visits at the clinical center. The total participation time is less than 24 hours.

Participants will have a medical interview and a neurological exam. They may give a urine sample before MRI.

Participants will have a short neuropsychologic and psychiatric interviews. Participants will have MRI scans. They will do small tasks or be asked to imagine things during the scanning.

DETAILED DESCRIPTION:
Eligibility:

DYT-SGCE patients and healthy volunteers (HV) between 15 and 60 years old.

ELIGIBILITY:
Inclusion Criteria:

For all participants:

* Age between 15-60 years
* Able to give informed consent.

For patients:

* An established diagnostic of DYT-SGCE
* No change in medication (related to DYT-SGCE) for a month

For controls:

* No neurological symptoms
* No medication except oral contraception

Exclusion Criteria:

* No deprivation of liberty
* Inability to give a consent
* Established cognitive alteration
* Contraindication to MRI (per MRI safety checklist)
* Severe chronic psychiatric illness

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The study will enroll patients with DYT-SGCE and Healthy Volunteers (HVs).
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2023-01-20 (Actual); Primary Completion 2024-02-19 (Actual); Study Completion 2024-02-19 (Actual)

PRIMARY OUTCOMES:
BOLD signal derived from the functional magnetic resonance imaging | 46 month
  Explore the differences in DYT-SGCE compared to HV

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Roze, Md, PhD, Principal Investigator — Department of neurology, Pitié-Salpêtrière Hospital, Paris
Locations (1):
- Brain Institute, Paris, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Roze E, Lang AE, Vidailhet M. Myoclonus-dystonia: classification, phenomenology, pathogenesis, and treatment. Curr Opin Neurol. 2018 Aug;31(4):484-490. doi: 10.1097/WCO.0000000000000577. PMID 29952836
- [Background] Peall KJ, Dijk JM, Saunders-Pullman R, Dreissen YE, van Loon I, Cath D, Kurian MA, Owen MJ, Foncke EM, Morris HR, Gasser T, Bressman S, Asmus F, Tijssen MA. Psychiatric disorders, myoclonus dystonia and SGCE: an international study. Ann Clin Transl Neurol. 2015 Nov 20;3(1):4-11. doi: 10.1002/acn3.263. eCollection 2016 Jan. PMID 26783545